CLINICAL TRIAL: NCT01785303
Title: Multidisciplinary Treatment for Obstructive Sleep Apnea and Insomnia
Brief Title: Multidisciplinary Approach to the Treatment of Insomnia and Comorbid Sleep Apnea
Acronym: MATRICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Stanford University (Other); National Jewish Health (Other); Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Jason Ong, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01HL114529-01 (NIH)
Record Dates: First submitted 2013-01-31; First posted 2013-02-07 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Obstructive Sleep Apnea; Insomnia
Keywords: CBT; CPAP; Multidisciplinary Treatment; Combination treatment
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Initiation and Maintenance Disorders | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Model A (Active Comparator): Model A consists of a 4 session CBT-I in phase I and CPAP for OSA in Phase II.
  Interventions: Behavioral: CBT-I; Procedure: CPAP
- Model B (Active Comparator): Model B consists of 4 weeks of monitoring using sleep diaries in Phase I. Phase II consists of concurrent initiation of CBT-I and CPAP for OSA.
  Interventions: Behavioral: CBT-I; Procedure: CPAP
- Model C (Other): Model C consists of 4 weeks of monitoring with sleep diaries in Phase I. Phase II consists of CPAP for OSA.
  Interventions: Procedure: CPAP

INTERVENTIONS:
Behavioral: CBT-I — Cognitive Behavior Therapy for Insomnia (CBT-I) consists of 4 weekly sessions delivered individually. The focus of these sessions is on modifying behaviors and cognitions related to sleep and insomnia.
  Other Names: CBT for Insomnia; CBT
  Arms: Model A; Model B
Procedure: CPAP — CPAP is an FDA-approved medical device used to treat obstructive sleep apnea. This device consists of a mask, hose, and machine that blows continuous air which maintains a consistent pressure of airflow preventing the upper airway from collapsing during sleep.
  Other Names: Continuous Positive Airway Pressure; Positive Airway Pressure

SUMMARY:
The overall goal of this project is to determine the efficacy of a multidisciplinary treatment model for patients with Obstructive Sleep Apnea (OSA) and comorbid Insomnia.

Specific Aim 1: To determine the efficacy of a treatment model combining Cognitive Behavioral Therapy (CBT) and Continued Positive Airway Pressure(CPAP) for individuals with OSA and comorbid insomnia.

Specific Aim 2: To determine if there are relative benefits in the sequence of treatment initiation.

Specific Aim 3: To examine the mechanisms between insomnia symptoms and CPAP adherence.

DETAILED DESCRIPTION:
OSA is a sleep-related breathing disorder that is growing in prevalence and is associated with negative cardiovascular consequences and adverse events from excessive daytime sleepiness. Insomnia is a frequently co-occurring sleep disorder that adds significant morbidity and is a potential barrier to adherence of OSA treatment. It is currently unknown if direct treatment of insomnia will enhance outcomes of OSA treatment. The investigators at the Rush Sleep Disorders Center have developed an approach that combines CBT for insomnia delivered by a psychologist with CPAP therapy managed by a physician. Building upon preliminary data collected in the clinic, the investigators seek to test the efficacy and mechanisms of this multidisciplinary model against the standard practice of treating OSA using CPAP alone.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females age 18 and older.
* Meets criteria for Obstructive Sleep Apnea
* Meets criteria for an Insomnia Disorder

Exclusion Criteria:

* Comorbid medical condition that requires immediate treatment of OSA
* Severe cases of OSA that require immediate treatment
* Psychiatric conditions that may interfere with study protocol or uncontrolled psychiatric conditions that require immediate treatment
* Comorbid sleep disorders that require treatment outside of the study protocol
* Other sleep-related breathing disorder besides OSA
* Excessive daytime sleepiness that requires immediate treatment or presents significant risk
* CPAP use or formal CBT for insomnia within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
CPAP adherence | 90 days after CPAP initiation
  CPAP adherence is defined as % nights used and hrs per night and % of "good users" (≥ 4 hours on ≥ 70% of nights)
Pittsburgh Sleep Quality Index (PSQI) | 90 days after CPAP initiation
  Improvements in sleep quality is defined as change of PSQI score from baseline to 90 days after CPAP initiation.

SECONDARY OUTCOMES:
Polysomnography (PSG) | End of phase 1 (1 month after baseline assessment)
  Improvement in PSG sleep efficiency at the end of Phase I
Insomnia Severity Index (ISI) | 90 days after CPAP initiation
  Improvement in ISI from baseline to 90 days after CPAP initiation
Functional Outcomes of Sleep Questionnaire (FOSQ) | 90 days after CPAP initiation
  Improvement in FOSQ from baseline to 90 days after CPAP initiation
Actigraphy | 90 days after CPAP initiation
  Improvement in sleep as measured by actigraphy from baseline to 90 days after CPAP initiation.

OTHER OUTCOMES:
Fatigue Severity Scale (FSS) | 90 days after CPAP initiation
  Improvement in FSS from baseline to 90 days after CPAP initiation (End of Phase II).
Epworth Sleepiness Scale (ESS) | 90 days after CPAP initiation
  Improvement in ESS from baseline to 90 days after CPAP initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Ong, PhD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Center for Circadian and Sleep Medicine, Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Turner AD, Ong JC, Jones AL, Tu A, Salanitro M, Crawford MR. Neurocognitive functioning in comorbid insomnia and sleep apnea patients is better after positive airway pressure therapy, but worse after cognitive behavioral therapy for insomnia: exploratory analysis of cognitive outcomes from the Multidisciplinary Approach to the Treatment of Insomnia and Comorbid Sleep Apnea study. Sleep. 2023 Aug 14;46(8):zsad128. doi: 10.1093/sleep/zsad128. PMID 37148183
- [Derived] Tu AY, Crawford MR, Dawson SC, Fogg LF, Turner AD, Wyatt JK, Crisostomo MI, Chhangani BS, Kushida CA, Edinger JD, Abbott SM, Malkani RG, Attarian HP, Zee PC, Ong JC. A randomized controlled trial of cognitive behavioral therapy for insomnia and PAP for obstructive sleep apnea and comorbid insomnia: effects on nocturnal sleep and daytime performance. J Clin Sleep Med. 2022 Mar 1;18(3):789-800. doi: 10.5664/jcsm.9696. PMID 34648425